CLINICAL TRIAL: NCT06808815
Title: A Phase I, Randomized, Double-Blinded, Placebo-Controlled, 3-Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending and Multiple Ascending Doses of S011806 in Healthy Participants and Multiple Doses of S011806 in Patients With Chronic Plaque Psoriasis
Brief Title: A Study to Assess S011806 (DC-806 or LY4100504) in Healthy Adult Participants and Participants With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DICE Therapeutics, Inc., a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCE806101; 2021-002888-21 (EudraCT Number); J5B-MC-FHAB (Other: Eli Lilly and Company); 297326 (Other: NHS Health Research Authority); 18850 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-01-31; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: DC-806 (Experimental): Single ascending dose of DC-806 administered orally.
  Interventions: Drug: DC-806
- Part 1: Placebo (Placebo Comparator): Placebo administered orally.
  Interventions: Other: Placebo
- Part 2: DC-806 (Experimental): Multiple ascending doses of DC-806 administered orally.
  Interventions: Drug: DC-806
- Part 2: Placebo (Placebo Comparator): Placebo administered orally
  Interventions: Other: Placebo
- Part 3:DC-806 (Experimental): DC-806 administered orally
  Interventions: Drug: DC-806
- Part 3: Placebo (Placebo Comparator): Placebo administered orally
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DC-806 — administered orally.
  Other Names: S011806; LY4100504
  Arms: Part 1: DC-806; Part 2: DC-806; Part 3:DC-806
Other: Placebo — administered orally.
  Arms: Part 1: Placebo; Part 2: Placebo; Part 3: Placebo

SUMMARY:
The main purpose of this study is to learn more about the safety and side effects of DC-806 when given by mouth to healthy participants and participants with Chronic Plaque Psoriasis. The study will have three parts. Each participant will enroll in only one part. For each participant, Part 1 will last up to 14 weeks, Part 2 will last up to 12 weeks, Part 3 will last up to 11 weeks including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects (Parts 1 and 2)

* Men and women participants must be between 18-55 years inclusive, at the time of informed consent.
* Female participants must either be of non-childbearing potential or if of childbearing potential, must not be pregnant, breast feeding or lactating and use a highly effective birth control method during treatment and for 90 days following last administered dose. In addition, male partners of female subjects of childbearing potential must use highly effective contraception for 90 days following the last administered dose
* Male participants who are sexually active with a partner of childbearing potential must use, with their partner, a condom plus an approved method of highly effective contraception from the time of informed consent until 90 days after their last dose of IMP.
* Participants must agree not to donate semen or ova/oocytes during the study and for 90 days after the last dose of IMP.
* Participants must have a body mass index (BMI) ≥ 18 and ≤ 35 kg/m2.
* Participants must be in good health as determined by medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory assessments at the time of screening, as judged by the Investigator or designee.

Participants with Psoriasis (Part 3)

* Men and women Participants must be between 18-65 years inclusive, at the time of informed consent.
* Participants must have a documented diagnosis of plaque psoriasis for ≥ 6 months prior to screening.
* Physicians Global Assessment (PGA) of 2/3 i.e. mild or moderate plaque psoriasis at baseline.
* Body Surface Area (BSA) ≥3% at baseline.
* A minimum of 2 psoriatic lesions of at least 2 cm x 2 cm at baseline, with at least 1 plaque in a site suitable for biopsy.
* Female participants must either be of non-childbearing potential or if of childbearing potential, must not be pregnant, breast feeding or lactating and use a highly effective birth control method during treatment and for 90 days following last administered dose. In addition, male partners of female subjects of childbearing potential must use highly effective contraception for 90 days following the last administered dose.
* Male participants who are sexually active with a partner of childbearing potential must use, with their partner, a condom plus an approved method of highly effective contraception from the time of informed consent until 90 days after their last dose of IMP.
* Participants must have a body mass index (BMI) ≥ 18 and ≤ 36 kg/m2.

Exclusion Criteria:

Healthy Subjects (Parts 1 and 2)

* History or presence of any clinically relevant acute or chronic medical or psychiatric condition that could interfere with the subject's safety during the clinical study or expose the subject to undue risk as judged by the Investigator or designee.
* After 10 minutes supine rest at the time of screening or prior to dosing on Day 1, any vital signs values outside the following ranges:

  * Systolic blood pressure <90 or >150 mmHg, or
  * Diastolic blood pressure <50 or >95 mmHg, or
  * Pulse <40 or >90 bpm
* Any clinically significant abnormalities in resting ECG at the time of screening or pre-dose Day 1 including prolonged QTcF (>450 ms for males; >470 ms for females using the mean of triplicate ECG's) and cardiac arrhythmias, as judged by the Investigator or designee.
* Clinically significant abnormalities in renal function:

  • eGFR <60 mL/min
* Clinically significant abnormalities in liver function:

  * Bilirubin >1.5 x ULN
  * Aminotransferases >1.5 x ULN
  * ALP >1.5 x ULN
* History of latent TB, active tuberculosis, or a positive QuantiFERON® TB Gold result at screening. Patients with an indeterminate QuantiFERON® TB Gold result at screening will be allowed one retest; if not negative on retesting, the subject will be excluded.
* Females who are pregnant, breast feeding or plan to be pregnant during the study period or 90 days after.
* Female subjects with a positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) at screening or within 24 h prior to the first administration of IMP.
* Positive serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCV Ab) or human immunodeficiency virus (HIV) 1 and/or 2 antibodies at screening.
* Part 2 Only: Presence of active suicidal ideation or positive suicide behaviour using the "Baseline/Screening" version of the Columbia Suicide Severity Rating Scale (C-SSRS) and with either of the following criteria:

  * History of a suicide attempt within the 5 years prior to the Screening Visit. Subjects with a history of a suicide attempt more than 5 years ago should be evaluated by a mental healthcare professional (eg, locally licensed psychiatrist, psychologist, or master's level therapist) before enrolling into the study.
  * Suicidal ideation in the past month prior to the Screening Visit as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Baseline/Screening" version of the C-SSRS.

Participants with Psoriasis (Part 3)

* History or presence of any clinically relevant acute or chronic medical or psychiatric condition other than psoriasis that could interfere with the patient's safety during the clinical study or expose the patient to undue risk as judged by the Investigator or designee.
* A diagnosis of non-plaque psoriasis.
* Plaque psoriasis restricted to the scalp, palms, soles and face.
* Pustular, erythrodermic, inverse, and guttate psoriasis
* Drug-induced psoriasis (i.e., new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium)
* Diagnosis of psoriatic arthritis, uveitis, inflammatory bowel disease, or other immune-mediated conditions that are commonly associated with psoriasis for which a subject requires current systemic (oral, SC, or IV) (including corticosteroids, immunosuppressants, biologics) immunosuppressant medical treatment
* Treatment with biologics within 5 half-lives (if known) or 6 months prior to dosing on Day 1, whichever is longer
* Has received any systemic immunosuppressants (e.g. Methotrexate, cyclosporine, hydroxyurea, and tacrolimus) or anakinra within 4 weeks of the first administration of study medication.
* Has received phototherapy or any systemic medications/treatments that could affect psoriasis or PGA evaluation (including, but not limited to, oral or injectable corticosteroids, retinoids, psoralens, sulfasalazine, hydroxyurea, apremilast, or fumaric acid derivatives) within 4 weeks of the first administration of study medication
* Has used topical medications/treatments that could affect psoriasis or PGA evaluation (including, but not limited to, corticosteroids, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, picrolimus, and tacrolimus) within 2 weeks of the first administration of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug. | Baseline Up To 7 Weeks
  A summary of AEs, TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the reported adverse events module.
Part 2: Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug. | Baseline Up To 7 Weeks
  A summary of AEs, TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the reported adverse events module.
Part 3: Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug. | Baseline Up To 11 Weeks
  A summary of AEs, TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the reported adverse events module.

SECONDARY OUTCOMES:
Part 1, Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of DC-806. | Pre-dose up-to 48 hours post-dose
  PK: Cmax of DC-806.
Part 1, PK: Area Under the Concentration Versus Time Curve (AUC) of DC-806. | Pre-dose up-to 48 hours post-dose
  PK: AUC of DC-806.
Part 1, PK: Time to reach maximum observed (Tmax) of DC-806 | Pre-dose up-to 48 hours post-dose
  PK: Tmax of DC-806
Part 1, PK: First-order elimination half-life (T1/2) of DC-806 | Pre-dose up-to 48 hours post-dose
  PK: Half-life (T1/2) DC-806
Part 2, PK: Maximum Observed Concentration (Cmax) of DC-806 | Pre-dose up-to 48 hours post-dose
  PK: Cmax of DC-806
Part 2, PK: Area Under the Concentration Versus Time Curve (AUC) of DC-806 | Pre-dose up-to 48 hours post-dose
  PK: AUC of DC-806
Part 2, PK: Time to reach maximum observed (Tmax) of DC-806 | Pre-dose up-to 48 hours post-dose
  PK: Tmax of DC-806
Part 2, PK: First-order elimination half-life (T1/2) of DC-806 | Pre-dose up-to 48 hours post-dose
  PK: Half-life (T1/2) DC-806
Part 3, PK: Maximum Observed Concentration (Cmax) of DC-806 | Pre-dose up-to 48 hours post-dose
  PK: Cmax of DC-806
Part 3, PK: Ctrough of DC-806 | Pre-dose up-to 48 hours post-dose
  pre-dose of DC-806

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 W Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- The Medicines Evaluation Unit (MEU) Ltd., Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No